CLINICAL TRIAL: NCT04328116
Title: Prospective Case Series Study of Neodent Implantable Devices of GM Zygomatic Line
Brief Title: Study of Neodent Implantable Devices of GM Zygomatic Line
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Other Study IDs: CS.O.008
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Jaw, Edentulous
Keywords: Dental Implants; Zygomatic Implants
MeSH Terms: conditions — Jaw, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Group: Neodent GM Zygomatic Dental Implants will be placed. Multiple implants may be placed in a single subject.
  Interventions: Device: Dental Implants

INTERVENTIONS:
Device: Dental Implants — Dental Implants will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the IFU (informations for use)

SUMMARY:
GM Zygomatic implant is intended to be surgically placed in the posterior region of the maxilla and zygoma. It is indicated for multiple prostheses in case of severe resorption in the maxilla and total edentulism (situations in which the installation of convectional implants is contraindicated).

The objective of the study is to confirm the long-term safety and clinical performance of GM Zygomatic implants and GM Zygomatic abutments in daily dental practice setting, by means of a prospective collection of clinical data concerning the success and survival rates of these devices.

Devices will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the instructions for use (IFU). Ten patients will be followed for 36 months and monitored for Adverse Events by the Investigators until the last protocol-related procedure of a patient is completed.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (CE) in Brazil.

GM Zygomatic implants present an optimized design with adapted treatment protocol, allowing for treatment of patients with severely resorbed maxilla and complete edentulism in which conventional implants placement is contraindicated.

The objective of the study is to confirm the long-term safety and clinical performance of implants and abutments of GM Zygomatic System in a daily dental practice setting, by means of a prospective collection of clinical data in a study using these devices.

Additionally, from the collected data, the study aims to identify previously unknown side-effects and monitor the known side-effects and contraindications stated on the Instructions for Use with the intent to verify that the intended purpose is adequate for all Neodent products involved in the procedure that come into contact with the patient.

The sample will be prospectively selected and will consist of 10 patients with atrophic edentulous maxillae, for whom the responsible surgeon elects the rehabilitation by means of placement of zygomatic implants as having the best risk-benefit ratio for the patient (e.g., shorter treatment time and lower biological cost than the associated with reconstructive surgeries for the insertion of conventional implants). Informed consent in writing will be obtained from each patient participating in the study prior to any study-related procedure.

Neodent GM Zygomatic implants will preferably be placed under local anesthesia and sedation (according to the surgeon's assessment of the patient's general health), with adequate bone bed preparation, as recommended by the manufacturer. Size, position, and quantity of implants (2 to 4) will be select considering the anatomy, region of rehabilitation, bone quality and quantity and available space. Together with the Zygomatic Implants, 2 to 4 conventional implants of Neodent GM line shall be inserted in the anterior region, if enough bone is available.

Data concerning the studied variables will be collected following the procedures and assessments plan by fulfilling the Case Report Form (CRF), in the following stages: First visit (Screening); T0 - Implants placement; TF - final prosthesis (may coincide with TL); TL - Implant loading; T6, T12, T24 and T36 - 6, 12, 24 and 36 months, respectively, after implant placement.

Computed tomography (CT) scans with prototyping will be obtained from the region of interest prior to surgery, for the surgical planning and implant selection, as well as post-surgery (T0 - immediately or within 1 week after implant placement; T36) to verify zygomatic implants anchorage. Prototypes of the region of interest in the maxilla will be obtained from the initial CT scans for diagnostic purposes. Additionally, standardized digital periapical radiographs will be taken in a usual daily practice frequency, as determined by the investigator: after implants placement (T0) and during the post-operative stages (TL, TF, T6, T12, T24, and T36) to assess the osseointegration process, changes in peri-implant bone level as well as prosthetic settlement and integrity.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more;
* Opposing dentition (natural teeth or teeth/implant-supported fixed restorations).

Exclusion Criteria:

* Symptomatology related to the facial sinuses (maxillary sinusitis, polyps or any other sinus pathologies);
* Unfavorable maxillary relations;
* Signs of allergy or hypersensitivity to the chemical ingredients of the material: titanium;
* Presence of acute inflammatory or infectious processes in live tissue;
* Unsuitable bone volume and/or quality;
* Systemic complications or diseases such as bone metabolism disorders, blood clotting disorders, unsuitable healing capacity, incomplete jawbone growth, uncooperative and not motivated patient, abuse of drugs or alcohol, psychosis, prolonged functional disorders which resist any treatment with medications, xerostomia, weakened immunological system, diseases which require the use of steroids, endocrine diseases, insufficient oral hygiene, and pregnancy.

Additionally, subjects will be excluded if they present systemic complications that may expose them to an eventual surgical risk if submitted to surgery under general anesthesia or under local anesthesia and sedation (decompensated diabetics, immunosuppressed, patients who were submitted to radiotherapy and chemotherapy less than 4 years or who had a heart attack less than 1 year previously, patients with clinical signs and/or symptoms of sinusitis and congestion and/or nasal secretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be prospectively selected and will consist of 10 patients with atrophic edentulous maxillae, for whom the responsible surgeon elects the rehabilitation by means of placement of zygomatic implants as having the best risk-benefit ratio for the patient (e.g., shorter treatment time and lower biological cost than the associated with reconstructive surgeries for the insertion of conventional implants).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | 36 months after implant placement.
  Implant survival will be defined as no loss of the implant at each follow-up.
Implant success rate | 36 months after implant placement.
  Evaluation of implant success will be assessed based on the criteria by Byser et al (1990).

SECONDARY OUTCOMES:
Implant survival rate | 6, 12, and 24 months after implant placement.
  Implant survival will be defined as no loss of the implant at each follow-up.
Implant success rate | 6, 12, and 24 months after implant placement.
  Evaluation of implant success will be assessed based on the criteria by Byser et al (1990).
Prosthetic survival rate | 12, 24, and 36 months after implant placement.
  Prosthetic survival will be assessed as the prosthesis remaining in situ at each follow-up, irrespective of its condition.
Prosthetic success rate | 12, 24, and 36 months after implant placement.
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention during the entire observational period.
Patient Satisfaction | Before implant placement and 6, 12, 24, and 36 months after implant placement.
  The portuguese translation of OHIP-14 [12,13] questionnaire will be used to assess Oral Health Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment.
Clinician Satisfaction | Immediately after implant placement, 12, 24, and 36 months after implant placement.
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction.
Adverse events related to the implant. | Immediately after implant placement, 6, 12, 24, and 36 months after implant placement.
  Determined by inquiring with the patient and clinical evaluation.
Adverse events related to the prosthesis. | Immediately after implant placement, 6, 12, 24, and 36 months after implant placement.
  Determined by inquiring with the patient and clinical evaluation.
Adverse events related to the surgery. | Immediately after implant placement, 6, 12, 24, and 36 months after implant placement.
  Determined by inquiring with the patient and clinical evaluation.
Adverse events related to the oral health | Immediately after implant placement, 6, 12, 24, and 36 months after implant placement.
  Determined by inquiring with the patient and clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Trojan, PhD, Study Chair — Neodent
Locations (1):
- Instituto Latino Americano de Pesquisa e Ensino Odontológico, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No